CLINICAL TRIAL: NCT04363970
Title: Early Versus Delayed Removal of the Urethral Catheter After Trans Urethral, Randomized Clinical Trial.
Brief Title: Early Removal of the Urethral Catheter Following Trans-urethral Resection of Prostate
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Saddam Al Demour, MD, University of Jordan
Other Study IDs: sad2020
Record Dates: First submitted 2020-04-16; First posted 2020-04-27 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Urinary Retention
Keywords: Benign Prostate Hyperplasia; Urinary retention; Re-catheterization
MeSH Terms: conditions — Urinary Retention; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A- early catheter removal): in group A, we will remove the catheter after 24 h.
  Interventions: Other: removal of the urinary catheter
- Group B- delayed catheter removal: In group B, we will remove the catheter after 48 h.
  Interventions: Other: removal of the urinary catheter

INTERVENTIONS:
Other: removal of the urinary catheter — in group A, we will remove the catheter after 24 h. In group B, we will remove the catheter after 48 h.

SUMMARY:
Transurethral resection of prostate is the gold standard operation for bladder outflow obstruction due to benign prostatic enlargement. However, catheter removal day is variable. The objective of this study is to compare early and delayed catheter removal groups in terms of, urinary retention after catheter removal, length of hospital stay, weight of resected prostate, duration of resection, peri-operative blood transfusion, and postoperative complications.

DETAILED DESCRIPTION:
This randomized controlled trial will carried out in Urology clinic at Jordan university hospital. Patients with benign prostate hyperplasia will be selected by simple random sampling technique after taking informed consent and will divided into two groups: Group A- early catheter removal group( catheter removed after 24 hours) and Group B-delayed catheter removal group ( catheter removed after 48 hours). in this study we will exclude patients with large post-void urine volume, simultaneous internal urethrotomy and transurethral resection of prostate, co-morbidity( diabetes mellitus, CVA) spinal cord injury, urethral stricture, prostate cancer proved by biopsy and intra-operative complications. Patients will discharged after removal of catheter if they voided successfully.

ELIGIBILITY:
Inclusion Criteria:

- All men with benign prostate hyperplasia who planned to undergo TURP will be included in this study.

Exclusion Criteria:

* Large post void residual urine.
* Simultaneous internal urethrotomy and TURP.
* Uncontrolled Diabetes Mellitus (DM).
* Cerebrovascular accident accident (CVA).
* Spinal cord injury.

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 adult males from urology clinic atJordan university hospital, with benign prostate hyperplasia who undergo trans-urethral resection of the prostae will be included in this study,
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
urinary retention | after 3 months.
  inability to void

SECONDARY OUTCOMES:
Lower urinary tract symptoms | after 3 months.
  urinary symptoms after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Saddam Al Demour, MD, Principal Investigator — Jordan University Hospital
Locations (1):
- Saddam Al Demour, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demour SA, Al-Zubi MT, Ababneh M, Al-Rawashdah SF, Ahmad M. A randomized clinical trial: timing of indwelling urethral catheter removal following transurethral resection of prostate. Future Sci OA. 2024 May 20;10(1):FSO927. doi: 10.2144/fsoa-2023-0195. eCollection 2024. PMID 38827798